CLINICAL TRIAL: NCT03669679
Title: Superomedial Pedicle Versus Inferior Pedicle in Breast Reduction Surgery
Brief Title: Comparison of Superomedial and Inferior Pedicle Techniques in Mammaplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed El-Sayed Sharaf Ahmed, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SM Vs Inf. Pedicle in BR
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Breast Hypertrophy
Keywords: breast reduction; mammaplasty; breast-q; patient satisfaction; patient reported outcome measures; superomedial pedicle; inferior pedicle
MeSH Terms: conditions — Gigantomastia; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): participants undergoing superomedial pedicle breast reduction "Hall-Findlay technique"
  Interventions: Procedure: Breast reduction
- Group B (Active Comparator): participants undergoing inferior pedicle breast reduction "Robbins technique"
  Interventions: Procedure: Breast reduction

INTERVENTIONS:
Procedure: Breast reduction — breast reduction surgery for breast hypertrophy using either superomedial or inferior pedicle technique

SUMMARY:
The aim of this study is to evaluate Superomedial pedicle and Inferior pedicle techniques in breast reduction for Egyptian females and compare between both pedicles regarding cosmetic outcomes, possible complications, patient satisfaction and time of operation.

DETAILED DESCRIPTION:
The female breast is one of the most attractive aesthetic areas in female anatomy. The size, shape, and symmetry of the breasts can have a dramatic effect on the women's wellbeing. Reduction mammaplasty is certainly one of the operations; plastic surgeons can significantly contribute to a woman's quality of life.

Macromastia or Breast Hypertrophy is a pathologic condition consisting of hypertrophy of the breast. It generates both physical and psychological distress, presenting a significant threat to a woman's health-related quality of life. Regarding Physical Distress Macromastia always associated with a number of musculoskeletal complications, including neck pain, back pain, headache, peripheral neuralgias, and shoulder pain. Often, women with mammary hypertrophy experience intertriginous skin maceration and other rashes, as well as infections all the result of heavy, pendulous breasts. In short, a woman's breast size can affect her attitudes, career choices, and personal life in many ways.

Ideal technique should end in a beautiful breast, which has good size with fullness in the upper part, attractive shape with adequate projection, elegant curves, and a nipple areola complex that is pleasing in shape and position. The result should last over years.

The inferior pedicle technique has been described with many variations by surgeons such as Ribeiro and Robbins with the nipple and areola being carried on a dermal pedicle, and it is probably one of the most popular breast reduction techniques currently in use in the United States. Advantages of this are well known. It is a rapid and safe technique that can be used on almost every breast size. It has been shown to be as good as or better than other techniques in the preservation of the neurovascular supply to the nipple. It is easily taught and learned.

The superomedial pedicle technique was first described by Orlando & Gutherie as a modification of the superior pedicle technique. In this technique the nipple & areola (NAC) is transposed on a superomedial de-epithelialized pedicle which contains a thin layer of subcutaneous tissue to protect the dermal blood supply.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral breast hypertrophy

Exclusion Criteria:

* Congenital breast anomalies.
* Pregnant, lactating or smoker patient.
* Previous breast reductions.
* Co-morbid diseases e.g. diabetes , liver cirrhosis or thyroid disorders.
* Body dysmorphic disorder
* Patients on long term medications e.g. immunosuppressive drugs, steroids or cytotoxic drugs.

Ages: 22 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 6 months
  evaluation of patient satisfaction pre/post-operatively using Arabic translated valid version of Breast-Q Reduction/Mastopexy Module (version 1)
Blood loss | 24 hours
  estimation of hemoglobin level deficit by evaluating hemoglobin level 24 hours post-operatively
Acute Complications | 2 weeks
  monitoring for the incidence of nipple & areola congestion/ischemia, hematoma, seroma, infection, wound dehisence or skin flaps congestion/ischemia
cosmetic outcomes | 6 months
  evaluation of breast symmetry, contour, projection, postoperative scars and shape of nipple & areola using standard photographs (anteroposterior, lateral and oblique views) by twoplastic surgery experts
Breast Measurements | 6 months
  * evaluation of breast vertical meridian and nipple to infra-mammary fold pre/post-operatively distance using tape measure
  * evaluation of breast degree of ptosis using Regnault's classification
Duration of the procedure | 6 hours
  estimation of the duration of the surgery from sterilization until application of the dressing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antony AK. Reply: A matched cohort study of superomedial pedicle vertical scar breast reduction (100 breasts) and traditional inferior pedicle wise-pattern reduction (100 breasts): an outcomes study over 3 years. Plast Reconstr Surg. 2014 Jun;133(6):885e-887e. doi: 10.1097/PRS.0000000000000210. No abstract available. PMID 24867750
- [Background] Ramon Y, Sharony Z, Moscona RA, Ullmann Y, Peled IJ. Evaluation and comparison of aesthetic results and patient satisfaction with bilateral breast reduction using the inferior pedicle and McKissock's vertical bipedicle dermal flap techniques. Plast Reconstr Surg. 2000 Aug;106(2):289-95; discussion 295-7. doi: 10.1097/00006534-200008000-00006. PMID 10946926
- [Background] Cabral IV, da Silva Garcia E, Sobrinho RN, Pinto NLL, Juliano Y, Veiga-Filho J, Ferreira LM, Veiga DF. Use of the BREAST-Q Survey in the Prospective Evaluation of Reduction Mammaplasty Outcomes. Aesthetic Plast Surg. 2018 Apr;42(2):388-395. doi: 10.1007/s00266-017-1009-6. Epub 2017 Nov 9. PMID 29124379